CLINICAL TRIAL: NCT00386425
Title: A Phase 2 Study to Evaluate Dose and Duration of Treatment of Drotrecogin Alfa (Activated) Using Serial Measurements of Protein C in Patients With Severe Sepsis and Multiple Organ Dysfunction
Brief Title: Evaluate Protein C Levels in Severe Sepsis Patients on Drotrecogin Alfa (Activated)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10553; F1K-MC-EVDK (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-11

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — drotrecogin alfa activated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard therapy (Experimental): 24 microgram/kilogram/hour (mcg/kg/hr) for 24 hours, followed by 24 mcg/kg/hr for an additional 72 hours
  Interventions: Drug: Drotrecogin alfa (activated)
- Alternative therapy:moderate protein C deficiency (Experimental): 24 mcg/kg/hr for 24 hours, followed by 24 mcg/kg/hr for an additional 48 to 144 hours (original protocol) or an additional 72 to 144 hours (amended protocol)
  Interventions: Drug: Drotrecogin alfa (activated)
- Alternative therapy:severe protein C deficiency (Experimental): 24 mcg/kg/hr for 24 hours, followed by 30 or 36 mcg/kg/hr for 48 to 144 hours (original protocol) or an additional 72 to 144 hours (amended protocol)
  Interventions: Drug: Drotrecogin alfa (activated)

INTERVENTIONS:
Drug: Drotrecogin alfa (activated) — intravenous
  Other Names: Xigris; LY203638

SUMMARY:
In this trial, patients with severe sepsis and low protein C levels will receive drotrecogin alfa (activated) at the normal, approved dose and time of administration [24 microgram/kilogram/hour (mcg/kg/hour) for 96 hours] or will receive the normal, approved dose or higher doses than the approved dose for a longer administration time. After the drug administration is complete, the protein C levels from the patients receiving the normal, approved dose will be compared to protein C levels from patients receiving the normal, approved dose or higher dose for a longer duration to determine if the protein C levels improve faster if given higher dose and/or longer administration time.

Note: The protocol was amended to remove the option of shorter infusion durations.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Must have a suspected or proven infection
* Must have two or more sepsis-associated organ dysfunctions

Exclusion Criteria:

* Documented multiple organ dysfunction greater than 24 hours prior to start of study drug
* Actual body weight less than 30 kg or more than 135 kg
* Platelet count less than 30,000/mm^3
* Active internal bleeding or at increased risk of bleeding
* Not expected to survive 28 days given the patient's pre-existing uncorrectable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2006-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (47):
- United States (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Loma Linda, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stanford, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abington, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
- Canada (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fleurimont, Quebec
- Finland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kuopio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oulu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampere
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Angoulême
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Roche-sur-Yon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Limoges
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tours
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell, Spain
- United Kingdom (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reading, Berkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brighton, East Sussex
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cottingham, East Yorkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kings Lynn, Norfolk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, West Midlands

REFERENCES:
- [Derived] Shorr AF, Janes JM, Artigas A, Tenhunen J, Wyncoll DL, Mercier E, Francois B, Vincent JL, Vangerow B, Heiselman D, Leishman AG, Zhu YE, Reinhart K; RESPOND investigators. Randomized trial evaluating serial protein C levels in severe sepsis patients treated with variable doses of drotrecogin alfa (activated). Crit Care. 2010;14(6):R229. doi: 10.1186/cc9382. Epub 2010 Dec 21. PMID 21176144

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Efficacy results are only provided for the intent-to-treat (ITT) population (patients who actually received the randomized treatment after the 24 hour pretreatment period).
Groups:
- Standard Therapy: 24 mcg/kg/hr for 24 hours, followed by 24 mcg/kg/hr for an additional 72 hours
- Alternative Therapy: Moderate Protein C Deficiency: 24 mcg/kg/hr for 24 hours, followed by 24 mcg/kg/hr for an additional 72 to 144 hours Severe Protein C Deficiency: 24 mcg/kg/hr for 24 hours, followed by 30 or 36 mcg/kg/hr for an additional 72 to 144 hours
- Randomized Non-ITT Population: Participants were randomized to either the Standard or Alternative Therapy and received 24 mcg/kg/hr during the first 24 hours (common therapy period); however, they did not continue on to receive the actual randomized therapy.
Period: Overall Study
Arm/Group | Standard Therapy | Alternative Therapy | Randomized Non-ITT Population
Started | 227 (51 severe protein C deficiency; 176 moderate protein C deficiency) | 206 (33 severe protein C deficiency; 173 moderate protein C deficiency) | 53
Received Study Drug | 227 | 206 | 53
Completed | 224 (51 severe protein C deficiency; 173 moderate protein C deficiency) | 205 (33 severe protein C deficiency; 172 moderate protein C deficiency) | 53
Not Completed | 3 | 1 | 0
Not completed — Physician Decision | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy | Alternative Therapy | Randomized Non-ITT Population | Total
Number analyzed (Participants) | 227 | 206 | 53 | 486
Age Continuous [Mean (Standard Deviation); unit: years] | 62.31 (16.11) | 61.91 (14.44) | 66.63 (12.82) | 62.61 (15.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 76 | 20 | 186
  Male | 137 | 130 | 33 | 300
Race/Ethnicity, Customized [Number; unit: Participants]
  African | 13 | 4 | 2 | 19
  Caucasian | 204 | 189 | 51 | 444
  East Asian | 0 | 2 | 0 | 2
  Hispanic | 9 | 8 | 0 | 17
  Native American | 0 | 1 | 0 | 1
  West Asian | 1 | 2 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Australia | 2 | 1 | 1 | 4
  Belgium | 27 | 23 | 6 | 56
  Canada | 22 | 21 | 4 | 47
  Germany | 14 | 12 | 1 | 27
  Finland | 29 | 30 | 2 | 61
  France | 37 | 33 | 9 | 79
  Italy | 1 | 1 | 0 | 2
  Puerto Rico | 2 | 4 | 0 | 6
  Spain | 19 | 16 | 12 | 47
  United Kingdom | 32 | 29 | 10 | 71
  United States | 42 | 36 | 8 | 86
Recent Surgery [Number; unit: participants] — Recent surgery was defined as an intervention performed under general or regional anesthesia that had some relationship to the present sepsis episode within 30 days of study entry.
  participants
    Yes | 68 | 61 | 25 | 154
    No | 159 | 144 | 28 | 331
    Unknown | 0 | 1 | 0 | 1
Number of organ dysfunctions [Mean (Standard Deviation); unit: organ dysfunctions] — Cardiovascular: systolic blood pressure (SBP) ≤90 mmHg or mean arterial pressure (MAP) ≤70 mmHg for >1 hour despite fluid resuscitation (FR), adequate intravascular volume, or vasopressors to maintain SBP ≥90 mmHg or MAP≥70 mmHg; Renal: average output <0.5 mL/kg/hr for 1 hr despite FR; Respiratory: Pressure of Arterial Oxygen (O2) to Fractional Inspired O2 (PaO2/FiO2) ≤250; Hematology: platelet count <80,000/mm^3 or 50% decrease in count from highest over 3 days prior to study; Unexplained acidosis: pH≤7.3 or base deficit ≥5.0 mEq/L AND plasma lactate level >1.5 times upper limit of normal.
  organ dysfunctions | 3.08 (0.86) | 3.08 (0.84) | 3.28 (0.93) | 3.10 (0.86)
Time of onset of Second organ dysfunction to start of drug infusion [Mean (Standard Deviation); unit: hours] — Mean time between the onset of a second organ dysfunction (cardiovascular, renal, respiratory, hematology, and unexplained metabolic acidosis) to the start of study drug infusion.
  hours | 15.3 (7.0) | 15.0 (7.0) | 15.8 (7.2) | 15.3 (7.0)
Total Sequential Organ Failure Assessment (SOFA) score [Mean (Standard Deviation); unit: units on a scale] — The presence of 5 organ dysfunctions (cardiovascular, respiratory, renal, hepatic, coagulation) was assessed using a Sequential Organ Failure Assessment (SOFA) score. Each organ has a possible dysfunction score of 0 to 4, for a total SOFA score range of 0 (no organ dysfunction) to 20 (all organs with dysfunction).
  units on a scale | 8.38 (2.83) | 8.65 (2.70) | 9.09 (2.25) | 8.57 (2.72)
Acute Physiology And Chronic Health Evaluation (APACHE) II Score [Mean (Standard Deviation); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation II. A classification system that assessed a patient's severity of disease based on 12 physiologic measurements, age, and previous health status. Total scores range from 0 to 71. A higher score indicates increasing severity of disease and a greater likelihood of mortality.
  units on a scale | 26.34 (7.70) | 26.15 (7.31) | 28.26 (8.05) | 26.47 (7.59)
Use of vasopressor [Number; unit: participants]
  Yes | 190 | 183 | 51 | 424
  No | 37 | 23 | 2 | 62
Mechanical ventilation [Number; unit: participants]
  Yes | 178 | 158 | 44 | 380
  No | 49 | 48 | 9 | 106
Protein C level [Mean (Standard Deviation); unit: Percent Protein C Activity] | 44 (19) | 41 (20) | 30 (18) | 42 (20)
Central laboratory protein C class [Number; unit: participants] — Moderate Protein C Deficiency: A protein C level greater than half the lower limit of normal.
  Severe Protein C Deficiency: A protein C level less than or equal to half the lower limit of normal.
  participants
    Severe deficiency | 97 | 100 | 31 | 228
    Moderate deficiency | 94 | 76 | 9 | 179
    Normal | 9 | 9 | 0 | 18
    Unknown | 27 | 21 | 13 | 61

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Protein C Levels From Day 1 to Day 7
Description: Mean change in protein C from Study Day 1 to Study Day 7 was tested using an unadjusted two-sample t-test with a two-sided alpha of 0.05. To be included in the primary analysis, Intention-to-Treat (ITT) patients must have at least 1 protein C value available at 24 hours or earlier and at least 1 protein C value at a post-24-hour timepoint.
Time Frame: Day 1, Day 7
Population: Intent to Treat (ITT) Last Observation Carried Forward (LOCF) population.
Measure: Mean (Standard Deviation); unit: Percent Protein C Activity
Arm/Group | Standard Therapy | Alternative Therapy
Number analyzed (Participants) | 227 | 206
Percent Protein C Activity
  Protein C Day 1, n=226, n=205 | 55 (24) | 52 (24)
  Protein C Day 7, n=221, n=203 | 79 (33) | 83 (35)
  Change in Protein C, Day 1 to Day 7, n=221, n=202 | 24 (29) | 31 (29)
Statistical Analysis 1: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.011, t-test, 2 sided — p-value is for change to Day 7

2. Secondary Outcome: Mean Change in Protein C Level From Study Day 1 to Study Day 7 in Patients With Moderate and Severe Protein C Deficiency
Description: Moderate Protein C Deficiency: A protein C level greater than half the lower limit of normal.
  Severe Protein C Deficiency: A protein C level less than or equal to half the lower limit of normal.
Time Frame: Day 1, Day 7
Population: ITT moderately deficient population, ITT severely deficient population
Measure: Mean (Standard Deviation); unit: Percent Protein C Activity
Arm/Group | Standard Therapy | Alternative Therapy
Number analyzed (Participants) | 227 | 206
Percent Protein C Activity
  Moderate n=175, n=171 | 24 (28) | 30 (29)
  Severe n=46, n=31 | 25 (32) | 38 (27)
Statistical Analysis 1: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.047, t-test, 2 sided — p-value is for the moderate Protein C Deficiency (difference in change of pc between alt and standard groups)
Statistical Analysis 2: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.063, t-test, 2 sided — p-value is for the severe Protein C Deficiency (difference in change of pc between alt and standard groups)

3. Secondary Outcome: Day 28 All-Cause Mortality
Time Frame: Day 0 through Day 28
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Standard Therapy | Alternative Therapy
Number analyzed (Participants) | 224 | 205
percentage of participants
  Alive at Day 28 | 83.9 | 75.1
  Deceased at Day 28 | 16.1 | 24.9
Statistical Analysis 1: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.030, Fisher Exact — p-value is for Day 28 mortality

4. Secondary Outcome: Hospital Mortality (up to Day 90)
Time Frame: Day 0 to hospital discharge or Day 90
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | Standard Therapy | Alternative Therapy
Number analyzed (Participants) | 224 | 205
Percentage of participants
  Discharged Alive | 79.5 | 72.2
  Deceased | 20.5 | 27.8
Statistical Analysis 1: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.090, Fisher Exact — p-value is for Day 90 mortality

5. Secondary Outcome: 28-Day Time Averaged Sequential Organ Failure (SOFA) Score
Description: The presence of 5 organ dysfunctions (cardiovascular, respiratory, renal, hepatic, coagulation) was assessed using a Sequential Organ Failure Assessment (SOFA) score. Each organ has a possible dysfunction score of 0 to 4, for a total SOFA score range of 0 (no organ dysfunction) to 20 (all organs with dysfunction). SOFA scores were time-averaged.
Time Frame: Day 0, Day 28
Population: ITT population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Standard Therapy | Alternative Therapy
Number analyzed (Participants) | 227 | 206
Units on a scale
  Total | 5.96 (5.21) | 6.62 (5.23)
  Cardiovascular | 1.28 (1.21) | 1.41 (1.26)
  Respiratory | 2.22 (0.99) | 2.38 (0.88)
  Renal | 0.92 (1.28) | 1.04 (1.31)
  Hematology | 0.80 (1.16) | 0.93 (1.20)
  Liver | 0.78 (1.22) | 0.89 (1.21)
Statistical Analysis 1: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.190, t-test, 2 sided — p-value is for total SOFA difference between alternative and standard therapy
Statistical Analysis 2: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.268, t-test, 2 sided — p-value is for difference in cardiovascular SOFA between alternative and standard therapy
Statistical Analysis 3: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.082, t-test, 2 sided — p-value is for difference in respiratory SOFA between alternative and standard therapy
Statistical Analysis 4: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.367, t-test, 2 sided — p-value is for difference in renal SOFA between alternative and standard therapy
Statistical Analysis 5: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.274, t-test, 2 sided — p-value is for difference in hematology SOFA between alternative and standard therapy
Statistical Analysis 6: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.341, t-test, 2 sided — p-value is for difference in liver SOFA between alternative and standard therapy

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) and Serious Bleeding Events (SBE) by Time Period
Description: Serious bleeding events (SBE): intracranial hemorrhage, life-threatening or fatal bleed, or bleeding event assessed as an SAE. Patients may have multiple events with onset in different time periods. SAEs include SBEs. The 3 SBEs in Alternative-Moderate Deficiency arm (days 5-8) occurred after completion of study drug infusion. One event (pleural haemorrhage) occurred same day of completion of infusion and 2 events (cerebral haemorrhage, shock haemorrhagic) occurred day after completion.
Time Frame: Day 0 through Day 28
Population: Randomized participants who received randomized therapy (intention to treat population).
Measure: Number; unit: number of patients with at least 1 event
Groups:
- Standard Therapy - Severe Deficiency; Standard Therapy - Moderate Deficiency: 24 mcg/kg/hr for 24 hours, followed by 24 mcg/kg/hr for an additional 72 hours
- Alternative Therapy - Severe Deficiency: Severe Protein C Deficiency: 24 mcg/kg/hr for 24 hours, followed by 30 or 36 mcg/kg/hr for an additional 72 to 144 hours
- Alternative Therapy - Moderate Deficiency: Moderate Protein C Deficiency: 24 mcg/kg/hr for 24 hours, followed by 24 mcg/kg/hr for an additional 72 to 144 hours
Arm/Group | Standard Therapy - Severe Deficiency | Standard Therapy - Moderate Deficiency | Alternative Therapy - Severe Deficiency | Alternative Therapy - Moderate Deficiency
Number analyzed (Participants) | 51 | 176 | 33 | 173
number of patients with at least 1 event
  Serious Bleeding Events: Study Days 0 through 4 | 0 | 2 | 0 | 9
  Serious Bleeding Events: Study Days 5 through 8 | 1 | 0 | 0 | 3
  Serious Bleeding Events: Study Days 9 through 28 | 0 | 1 | 0 | 1
  Serious Adverse Events: Study Days 0 through 4 | 0 | 10 | 5 | 17
  Serious Adverse Events: Study Days 5 through 8 | 2 | 4 | 1 | 8
  Serious Adverse Events: Study Days 9 through 28 | 3 | 8 | 4 | 14

7. Secondary Outcome: Mortality by Protein C Normalized Versus Not-normalized
Description: Normalization was defined as having 2 consecutive protein C measurements above the lower limit of normal through Study Day 7.
Time Frame: 28 days
Population: ITT Population - All patients who are randomly assigned to treatment and receive any amount of randomized therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Normalized Protein C | Did Not Normalize Protein C
Number analyzed (Participants) | 232 | 197
Percentage of participants | 10.3 | 32.0
Statistical Analysis 1: Comparison: Normalized Protein C vs Did Not Normalize Protein C; Test type: Superiority or Other; p < 0.0001, Fisher Exact — p-value is for difference between participants normalizing protein C and not normalizing protein C

8. Other Pre Specified Outcome: Mortality for Severe Protein C Deficiency
Description: Twenty-eight day mortality is the patient's mortality status at the predefined timepoint of 672 hours from the start of study drug infusion. Hospital mortality is the patient's survival status at the end of the hospital stay or study day 90 (if the patient remains in the hospital).
Time Frame: 28 Days, up to 90 days
Population: ITT Population - All patients who are randomly assigned to treatment and receive any amount of randomized therapy. ITT patients with severe protein C deficiency. Severe deficiency is defined by the 24-hour local laboratory protein C value reported to the Interactive voice response system (IVRS).
Measure: Number; unit: Percentage of participants
Arm/Group | Standard Therapy | Alternative Therapy
Number analyzed (Participants) | 51 | 33
Percentage of participants
  28 Day Mortality - Deceased at Day 28 | 31.4 | 24.2
  28 Day Mortality - Alive at Day 28 | 68.6 | 75.8
  Hospital Mortality - Deceased | 33.3 | 30.3
  Hospital Mortality - Discharged Alive | 66.7 | 69.7
Statistical Analysis 1: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.622, Pearson's chi-square test — p-value is for 28-Day Mortality, Dead at Day 28 vs. Alive at Day 28
Statistical Analysis 2: Comparison: Standard Therapy vs Alternative Therapy; Test type: Superiority or Other; p = 0.815, Fisher Exact — p-value is for Hospital Mortality

9. Post Hoc Outcome: Mortality for Moderate Protein C Deficiency by Infusion Duration
Time Frame: 28 Days
Population: ITT Population - ITT Switch-No Population, ITT patients who did not answer yes to the switch question.
Measure: Number; unit: percent participants deceased
Arm/Group | Standard Therapy | Alternative Therapy
Number analyzed (Participants) | 135 | 142
percent participants deceased
  <97 Hours n=65, n=71 | 13.8 | 28.2
  >=97 Hours n=70, n=71 | 11.4 | 23.9

ADVERSE EVENTS:
Groups:
- Standard Therapy: Participants assigned to standard therapy (24 mcg/kg/hr for 24 hours, followed by 24 mcg/kg/hr for an additional 72 hours) who received any amount of study drug.
- Alternative Therapy: Participants assigned to alternative therapy (Moderate Protein C Deficiency: 24 mcg/kg/hr for 24 hours, followed by 24 mcg/kg/hr for an additional 72 to 144 hours Severe Protein C Deficiency: 24 mcg/kg/hr for 24 hours, followed by 30 or 36 mcg/kg/hr for an additional 72 to 144 hours) who received any amount of study drug.
Arm/Group | Standard Therapy | Alternative Therapy
Serious Adverse Events (participants affected / at risk) | 33/250 | 48/236
Other Adverse Events (participants affected / at risk) | 51/250 | 46/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=250) | Alternative Therapy (N=236)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Electromechanical dissociation (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 1 (1)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Candida pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 4 (4)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 2 (2)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Therapy (N=250) | Alternative Therapy (N=236)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 1 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloody discharge (General disorders) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 4 (6) | 5 (9)
Mucosal haemorrhage (General disorders) | 2 (2) | 2 (2)
Puncture site haemorrhage (General disorders) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 2 (2)
Catheter sepsis (Infections and infestations) | 2 (2) | 1 (1)
Citrobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Morganella infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 3 (3) | 2 (2)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Bloody airway discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Bacteria blood identified (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Prothrombin time shortened (Investigations) | 0 (0) | 2 (2)
Sputum culture positive (Investigations) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 3 (3) | 1 (1)
Wound haemorrhage (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Fewer patients than planned had severe PC deficiency so only 2 higher doses were tested & fewer required longer infusions so a large proportion of alternative therapy patients in effect received standard therapy making treatment comparisons difficult

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days